CLINICAL TRIAL: NCT03531138
Title: Is it Possible to Use the Timed Performance Tests in Lung Transplantation Candidates to Determine the Exercise Capacity?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Principal investigator, Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: performans_2018
Record Dates: First submitted 2018-05-09; First posted 2018-05-21 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Pulmonary Rehabilitation; Exercise Capacity; Exercise Test
Keywords: performance test; exercise capacity; rehabilitation outcome; pulmonary rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary rehabilitation group (Experimental): All patients will undergo supervised pulmonary rehabilitation program on 2 days per week for 3 months. Apart from that, they will ask to perform the home exercise program which is scheduled as 3 days per week.
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Pulmonary Rehabilitation — All patients will undergo supervised pulmonary rehabilitation program on 2 days per week for 3 months. Apart from that, they will ask to perform the home exercise program which is scheduled as 3 days per week and fill out the exercise follow-up form. Supervised exercise sessions consist of aerobic(treadmill walking, bicycle training, arm ergometer training) and strengthening training(free weights). A 6-min walk test, a 10-meter walking speed test and a 5 times sit to stand test will be performed to determine the exercise capacity of the patient. The tests will be carried out at the beginning and end of rehabilitation. At each testing session, the tests will be performed sequentially by the same physiotherapist, giving 20 minute rest periods within the same day.

SUMMARY:
Lung transplantation candidates will be performed a 3-month hospital-based preoperative exercise training. A 6-minute walk test, a 10-meter walking speed test and a 5-times sit to stand test will be performed to determine the exercise capacity of the patient. The tests will be carried out at the beginning and end of rehabilitation. At each testing session, the tests will be performed sequentially by the same physiotherapist, giving 20 minute rest periods within the same day. It will be analyzed how the test data correlate with each other and how the delta values calculated for each test reflect the rehabilitation outcomes calculated after the exercise program.

DETAILED DESCRIPTION:
Severe exercise intolerance exists in lung transplant candidates. Completion of the test period in the field tests used in determining the exercise capacity of these patients is extremely difficult. The exercise capacity, which is considered as an important criterion in the decision of the lung transplant decision and in the determination of the clinical profile of the patient, necessitates the development of different test methods which are more suitable for the application of the measurement in this patient population.

In this study lung transplantation candidates will be performed a 3-month hospital-based preoperative exercise training. A 6-minute walk test, a 10-meter walking speed test and a 5-times sit to stand test will be performed to determine the exercise capacity of the patient. The tests will be carried out at the beginning and end of rehabilitation. At each testing session, the tests will be performed sequentially by the same physiotherapist, giving 20 minute rest periods within the same day. It will be analyzed how the test data correlate with each other and how the delta values calculated for each test reflect the rehabilitation outcomes calculated after the exercise program.

ELIGIBILITY:
Inclusion Criteria:

* To be taken to the list for lung transplant
* Do not have any addiction that may interfere with exercise

Exclusion Criteria:

-Do not accept to study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline distance covered in six minute walking test at 3-months | 3-months
  The test was conducted in a 30-meter corridor in line with American Thoracic Society (ATS) guidelines. Patients were told that they should walk as fast as they can walk. Before and after the test, oxygen saturation, heart rate, Borg fatigue rating, and walking distance were recorded.
Change from baseline 10-meter walking speed test at 3-months | 3-months
  The patient walks without assistance 10 meters (32.8 feet) and the time is measured.
Change from baseline 5 times sit to stand test at 3-months | 3-months
  Patient stand up and sit as quickly as possible from a standard chair for 5 times.Introduction: "Stand up and sit down as quickly as possible 5times, keeping your arms folded across your chest. I'll be timing you with a stopwatch. Ready, begin".The time is measured. Lower times = better scores.

SECONDARY OUTCOMES:
Change from baseline Modified Medical Research Council (mMRC) Dyspnea Scale score at 3-months | 3-months
  The mMRC Dyspnea Scale is best used to establish baseline functional impairment due to dyspnea attributable to respiratory disease; tracking the mMRC over time or with therapeutic interventions is of less certain clinical utility.The severity of dyspnea is rated on a scale of 0 to 4. "O" means no dyspnea perception, "4" means severe dyspnea perception.
Change from baseline Maximum Inspiratory Pressure (MIP) at 3-months | 3-months
  The mouth pressure measurement was performed with the Micro-RPM® instrument from SensorMEDIC. Patient placed a rubber mouthpiece with flanges, on the device, sealed their lips firmly around the mouthpiece, exhaled/inhaled slowly and completely, and then tried to breath in as hard as possible. The patient was allowed to rest for about a minute and the maneuver was repeated five times. Verbal or visual feedback was provided after each maneuver. The aim is that the variability between measurements is less than 10 cm H2O. The maximum value was obtained.
Change from baseline Forced Expiratory Volume in 1 second (FEV1) at 3-months. | 3-months
  It was conducted by using the Sensor Medics model 2400 (Yorba Linda, CA, USA), and according to the American Thoracic Society (ATS) guidelines.
Change from baseline quadriceps femoris muscle strength at 3-months. | 3-months
  Muscle Strength will measure using a digital dynamometer (J-Tech Commander muscle testing device), wth three measurements make. Best result will be taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Yedikule Chest Disease Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided